CLINICAL TRIAL: NCT07028814
Title: Risk Informed Obesity Care Plan Pilot
Status: Enrolling by invitation | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief Community Health & Health Equity Officer, Massachusetts General Hospital
Other Study IDs: 2025P001605
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Risk-informed obesity care plan: Children aged 2-12 years with overweight or obesity receiving primary care from a participating provider
  Interventions: Other: Risk-informed obesity care plan

INTERVENTIONS:
Other: Risk-informed obesity care plan — A risk-informed obesity care plan, implemented through pediatric primary care provider training via a Virtual Learning Collaborative (VLC) will be deployed.

SUMMARY:
The purpose of this research is to conduct a pilot of a risk-informed obesity care plan, implemented through pediatric primary care provider training via a Virtual Learning Collaborative (VLC) at MGH's Healthy Weight Clinic. We will evaluate HEDIS documentation and BMI outcomes among kids who receive care from the participating providers during and after the training period, compared to those who received care from the providers prior to the training.

ELIGIBILITY:
Inclusion Criteria:

* Child 2-12 years of age at baseline
* Child has overweight or obesity, based on their height/weight measurement
* Child presented for primary care with a medical provider participating in the training

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be patients of medical providers participating in the MGH Healthy Weight Clinic and Asthma Control Program's Virtual Learning Community
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
HEDIS documentation codes | 0-6 months

SECONDARY OUTCOMES:
Change in child Body Mass Index from baseline to 6 months | 0-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This retrospective data pull will be used for the evaluation of our aims, and is purposefully limited to only the required information. Interest parties can contact the PI to request IPD and the rationale for consideration on a case by case basis.